CLINICAL TRIAL: NCT03298607
Title: The Impact of Sérélys PMS, a Herbal Remedy Based on Pollen Extraction and Saffron, on Symptoms of PMS: A Randomized, Double-blinded, Placebo Controlled Study
Brief Title: The Impact of Serelys PMS on Symptoms of PMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Serelys Pharma (Unknown)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Adj Professor, Department of Nutrition, Exercise and Sports, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-17014613
Record Dates: First submitted 2017-09-07; First posted 2017-10-02 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: 2 months treatment with (Food Supplement - Serelys PMS)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2 capsules daily for 2 months containing inactive substances
  Interventions: Dietary Supplement: Placebo
- Serelys PMS (Active Comparator): 2 capsules daily for 2 months containing pollen extract
  Interventions: Dietary Supplement: Serelys PMS

INTERVENTIONS:
Dietary Supplement: Placebo — 2 months treatment
  Arms: Placebo
Dietary Supplement: Serelys PMS — 2 months treatment
  Arms: Serelys PMS

SUMMARY:
The objective of the present study is to better define and evaluate Serelys PMS in terms of the impact on the different premenstrual syndrome (PMS) symptoms , tolerance, satisfaction and overall quality of life of women with known discomforts during the premenstrual period. The data from this study will be compared to data when the two different ingredients are given as monotherapy.

DETAILED DESCRIPTION:
More than every other women aged 15 to 50 years of age have premenstrual symptoms such as irritability, mood swings, fatigue, headaches, sleep disturbances, breast and abdominal pain, bloating, water retention and weight gain. Some signs continue during menstruation. These psychological and physical manifestations can make women vulnerable and have a negative impact on their professional, social and sexual life. Randomized, double-blind, placebo-controlled clinical studies demonstrated the beneficial effects of pollen extract in premenstrual discomfort. The premenstrual period is probably caused by a change in the normal amount of sex hormones which can induce disorders in the central neuroendocrine system and estrogens are reported to reduce PMS symptoms to some extend. Moreover, it is well established that serotonin may play a role in PMS, as some inhibitors of serotonin re-uptake (SSRI) have an impact on premenstrual disorders. However, side effects may occur even when using estrogens as well as SSRI. Recently the pollen extract formulation has been improved by adding a natural extract of saffron. This latter component is known for its beneficial action on maintaining comfort during the menstrual cycle of the woman and it especially supports mood changes, one of the mayor PMS symptoms. The effect of Safran was studied more specifically in a randomized controlled double-blind, placebo-controlled clinical trial in women with premenstrual discomfort. This study showed a progressive and significant improvement after the use of saffron. In an other study saffron was documented to improve mood in patients with milder depression.

In summary, the components of saffron helps to improve the well-being of women during the premenstrual and menstrual period and have a well documented impact on mood. The pollen based extracts have well documented impact on most of PMS symptoms but possibly lesser on mood changes, which is also one of the mayor symptoms of PMS. The mechanisms by which saffron and pollen based extraction works is expected to be different and an additive impact is expected. The investigation is initiated by the researchers who feel that in PMS an alternatives to SSRI and estrogen treatment is needed.

ELIGIBILITY:
Inclusion Criteria:

* At least five inconveniences in the premenstrual period and which disappear quickly with the end of menstruation : Irritability, Tension, Fatigue, Dysphoria (sadness), Reduced motor coordination, Difficulty concentrating, Changes in libido, Changes in appetite.
* these inconveniences disappear quickly with the end of menstruation
* At least one of these criteria must be present in the premenstrual and menstrual period:

  1. Deterioration in relations with the family, at home, in school or at work
  2. Having thought to take painkillers for at least one menstrual cycle.
* Have symptoms of dysphoria / premenstrual sadness at least during the previous 6 cycles.

Exclusion Criteria:

* Known allergy to any component of the product and known renal and hepatic impairment.
* Existence of major evolving pathologies
* Convulsions. Existence of psychiatric disorders, cravings
* Suicidal thoughts
* Taking medications that may interfere with PMS symptoms like eg estrogens.
* Participation in another clinical study at the same time.
* Pregnancy and / or lactation;
* Difficulties to collaborate and difficulties to understand and complete the questionnaires.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
PMS symptoms evaluation - Premenstrual Tension | 2 months
  Premenstrual Tension Scale (PMTS) - Self-rating scale
PMS symptoms evaluation - Premenstrual Tension 2 | 2 months
  Premenstrual Tension Scale (PMTS) - Observe Rating Scale
PMS symptoms evaluation - premenstrual discomfort | 2 months
  Evaluation of premenstrual discomfort by Visual Analog Scales (VAS)

SECONDARY OUTCOMES:
Side effect registration | 2 months
  Tolerance will be assessed through a scoring system
Satisfaction scored by the patients | 2 months
  Satisfaction and well-being will be assessed through a scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Winther Hansen, MD, Study Chair — UCopenhagen, Department of Nutrition, Exercise and Sport
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No